CLINICAL TRIAL: NCT06065436
Title: Impact of Concurrent Low Intensity Shockwave Therapy on Clinical Outcomes With Collagenase Clostridium Histolyticum in Peyronie's Disease: A Randomized Controlled Trial
Brief Title: Concurrent Low Intensity Shockwave Therapy on Collagenase Clostridium Histolyticum for Peyronie's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tobias S. Kohler, MD, MPH, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-002478
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Peyronie Disease; Erectile Dysfunction
MeSH Terms: conditions — Penile Induration; Erectile Dysfunction | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Collagenase Clostridium Histolyticum with Low Intensity Shockwave Therapy (Experimental): Subjects will receive Collagenase Clostridium Histolyticum (CCH) intralesional injection with low-intensity shockwave therapy (LiSWT).
  Interventions: Drug: Collagenase Clostridium Histolyticum; Device: Storz Duolith LiSWT
- Collagenase Clostridium Histolyticum (Active Comparator): Subjects will receive Collagenase Clostridium Histolyticum (CCH) intralesional injection per standard of care.
  Interventions: Drug: Collagenase Clostridium Histolyticum

INTERVENTIONS:
Drug: Collagenase Clostridium Histolyticum — Total of 8 Intralesional injection (0.90 mg), administered as four separate injection series. Within each series, subjects will receive two injections, administered approximately 1-7 days apart.
  Other Names: Xiaflex
Device: Storz Duolith LiSWT — Single low intensity shockwave therapy consistent of 1,500 shocks at a rate of 120 shocks/minute and using a power setting of 0.09 mJ/mm2. These treatments will occur four separate times, before each of the four separate CCH injection series.
  Arms: Collagenase Clostridium Histolyticum with Low Intensity Shockwave Therapy

SUMMARY:
The purpose of this research is to determine whether or not low-intensity shockwave therapy (LiSWT) with Xiaflex treatment will result in greater improvements to the curvature of the penis.

ELIGIBILITY:
Inclusion Criteria

• Diagnosed with PD

* Palpable penile plaque
* Dorsal, lateral, or dorsolateral penile curvature
* Penile curvature > 30 degrees and < 90 degrees as measured using goniometer during objective curvature assessment
* Non-calcified plaque or grade 1 calcification ("stippling", no shadowing) as determined by penile duplex Doppler ultrasound (PDDU)
* "Stable PD symptoms' defined as PD symptom duration > 6-months or stable symptoms > 3-months

Exclusion Criteria:

* Prior intralesional injections or surgery for PD.
* Severe baseline penile pain.
* Moderate or severe baseline ED based on IIEF-EF domain.
* History of low intensity shockwave therapy for sexual dysfunction (ED or PD).
* Ventral (downward) or ventrolateral penile curvature.
* Moderate or severe (grade 2/3) plaque calcification as determined by PDDU.
* Inability to achieve satisfactory erection rigidity at time of baseline curvature assessment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in symptom bother | Baseline, 6 weeks
  Measured using the validated Peyronie's Disease Questionnaire (PDQ) subdomain symptom bother. Four questions to evaluate pain or discomfort during vaginal intercourse: responses include "not at all bothered", "a little bit bothered" , "moderately bothered", "very bothered", "extremely bothered"
Change in penetrative sexual intercourse | Baseline, 6 weeks
  Measured using self-reported question: "Over the past 4 weeks: When you attempted intercourse, how often were you able to penetrate (enter) your partner?" Responses include "no sexual activity", "almost never or never" , "a few times (less than half the time)", "sometimes (about half the time)", "Most times (more than half the time)", "almost always or always.
Surgical straightening intervention | 6 weeks
  Number of subjects to require surgical straightening
Change in erectile function | Baseline, 6 weeks
  Measured using the International Index of erectile Function
Change in Erectile Function Domain (IIEF-EF) | Baseline, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kohler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20556913#overview